CLINICAL TRIAL: NCT06365450
Title: OWEL Cancer Education and Awareness Program (OCEAP)
Brief Title: Breast and Cervical Cancer Education Program
Acronym: OCEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Older Women Embracing Life (Unknown); The John G. Bartlett Specialty Practice (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00315481
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer; Breast Cancer; Health Behavior
MeSH Terms: conditions — Uterine Cervical Neoplasms; Breast Neoplasms; Health Behavior | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Each participant is required to attend (in person or virtually via Zoom) two educational sessions one on breast cancer and the other on cervical cancer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Single-group (Experimental): 1 educational session on cervical cancer and one educational session on breast cancer
  Interventions: Other: Educational Intervention

INTERVENTIONS:
Other: Educational Intervention — Participants will receive hybrid educational intervention on breast and cervical cancer

SUMMARY:
The primary goal of this study is to improve cancer literacy in Black women living with HIV and ultimately improve breast and cervical cancer screening uptake. This study involves an educational intervention delivered virtually and in person, depending on the participants' preference.

DETAILED DESCRIPTION:
The aims of this study are to:

1. develop educational materials on breast and cervical cancer screening;
2. administer the intervention using a PowerPoint presentation;
3. evaluate changes in breast and cervical cancer literacy levels after the intervention; and
4. assess participants'; satisfaction with the program

ELIGIBILITY:
Inclusion Criteria:

* able to read and write in English
* self-identify as HIV positive -
* Black/African American.

Exclusion Criteria:

* Acutely ill

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Health Literacy in Cancer Screening as assessed by the Assessment of Health Literacy in Cancer Screening (AHL-C) tool. | Immediately Post intervention
  The dimensions of health literacy adapted from the AHL-C tool are:
  1. Numeracy (2 items)
  2. Familiarity (9 items)
  3. Comprehension (1 item)
  4. Navigation (7 items).
  To determine health literacy scores of participants, each item will be scored on a scale of 0 to 1. A higher score would mean a better outcome. Items will be summed for each of the four sub-scales as well as the entire scale (AHL-C) and then determine the mean and standard deviation.
  Assessment will be completed immediately post intervention (after two sessions on breast and cervical cancer)

SECONDARY OUTCOMES:
Number of participants recruited from each community partner | Immediately Post intervention
  Participants recruited from each community partner
Number of participants who preferred virtual or in person sessions | Immediately Post intervention
  Participant session attendance preference
Number of participants who were lost of follow up | Immediately post intervention
  Participants lost to follow up
Number of participants who needed help redeeming their gift codes | Immediately post intervention
  Participants needing help redeeming gift cards

CONTACTS AND LOCATIONS:
Overall Officials: Hae-Ra Han, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No